CLINICAL TRIAL: NCT07220538
Title: Pragmatic Open-label, Parallel-group Clinical Trial on the Effectiveness of Extract of Ginkgo Biloba Leaves Tablets as add-on to Standard of Care in Participants With Cognitive Impairment After an Acute Ischemic Stroke (GiCIIS)
Brief Title: A Study Testing How Well the Drug Extract of Ginkgo Biloba Leaves Tablets Works for People With Memory or Thinking Problems After a Stroke When Added to Standard Treatment
Acronym: GiCIIS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Dr. Willmar Schwabe GmbH & Co. KG (Industry)
Collaborators: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D.01.02.2.04; ChiCTR2500107051 (Registry Identifier: China Clinical Trial Registry)
Record Dates: First submitted 2025-10-14; First posted 2025-10-24 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-11

CONDITIONS: Ischemic Stroke Hospitalized; Impairment, Cognitive
Keywords: Acute ischemic stroke; Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction; Ischemic Stroke | interventions — Standard of Care; Population Groups

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extract of Ginkgo Biloba Leaves Tablets 240 mg (2 x 40 mg, t.i.d.) add-on to standard of care (Experimental): Extract of Ginkgo Biloba Leaves Tablets 240 mg (2 x 40 mg, t.i.d.) add-on to standard of care
  Interventions: Drug: Extract of Ginkgo Biloba Leaves Tablets 240 mg (2 x 40 mg, t.i.d.)
- Standard of Care (Sham Comparator): Standard of Care (SoC) Group
  Interventions: Other: Standard of care (SoC) Group

INTERVENTIONS:
Drug: Extract of Ginkgo Biloba Leaves Tablets 240 mg (2 x 40 mg, t.i.d.) — 3 x 2 film-coated tablets with 40 mg Extract of Ginkgo Biloba Leaves Tablets daily for 52 weeks plus standard of care in accordance with treatment guidelines
  Arms: Extract of Ginkgo Biloba Leaves Tablets 240 mg (2 x 40 mg, t.i.d.) add-on to standard of care
Other: Standard of care (SoC) Group — Individualized therapy in accordance with treatment guideline from the Chinese Stroke Association
  Arms: Standard of Care

SUMMARY:
The goal of this clinical trial is to learn if Extract of Ginkgo Biloba Leaves Tablets help improve thinking and memory in people aged 55 years and older who had an ischemic stroke (a type of stroke caused by a blocked blood vessel in the brain). It will also look at how safe the Extract of Ginkgo Biloba Leaves Tablets are.

The main questions it aims to answer are:

* Do the Extract of Ginkgo Biloba Leaves Tablets help people with memory or thinking problems after an ischemic stroke?
* What medical problems do people have when taking the Extract of Ginkgo Biloba Leaves Tablets ? Researchers will compare people who take the Extract of Ginkgo Biloba Leaves Tablets along with their usual post-stroke treatment to people who only receive their usual post-stroke treatment.

Participants will:

* Have had an ischemic stroke confirmed by MRI (Magnet Resonance Imaging, a magnetic scan that helps seeing inside the body in great detail) 7 to 14 days before joining the study
* Take Extract of Ginkgo Biloba Leaves Tablets (240 mg per day) in addition to usual post-stroke treatment for 12 months, or receive only usual post-stroke treatment for 12 months
* Be treated initially at hospitals across China
* Visit the clinic 4, 26, and 52 weeks following the baseline for checkups and tests, and receive follow-up calls after 12 and 38 weeks.

DETAILED DESCRIPTION:
This is a prospective, multicenter, pragmatic, open-label, parallel-group, randomized clinical trial to investigate the effectiveness and safety of Extract of Ginkgo Biloba Leaves Tablets as add-on to standard of care in participants with cognitive impairment after an acute ischemic stroke (AIS). The trial will be conducted at hospitals across China. Participants that had had a non-disabling overt AIS (i. e., NIHSS (National Institutes of Health Stroke Scale) ≤ 5, mRS (Modified Rankin Scale) ≤ 2 at the day of screening), confirmed by MRI (magnetic resonance imaging), 7 to 14 days before screening will be randomized 1:1 to Extract of Ginkgo Biloba Leaves Tablets (240 mg total dose per day, (3 x (2 x 40 mg)) in addition to standard of care or standard of care alone. The total duration of the trial will be 52 weeks per trial participant.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants aged ≥ 55 years who gave their informed consent.
2. Non-disabling overt acute ischemic stroke (NIHSS (National Institutes of Health Stroke Scale) ≤ 5, mRS (Modified Rankin Scale) ≤ 2 at the day of screening) confirmed by magnetic resonance imaging, and at least 7 but no longer than 14 days before baseline.
3. Cognitive impairment (MoCA (Montreal Cognitive Assessment)) total score (corrected) < 23 for participants with up to 12 years of education, or MoCA total score < 22 if more than 12 years of education).
4. Sufficient Chinese language skills to understand and respond to all interview questions, complete questionnaires and undergo neuropsychological testing.

Exclusion Criteria:

1. Participation in another experimental drug trial at the same time or within the past 4 weeks before enrollment.
2. Aphasia, dysarthria, apraxia or paresis of the dominant upper extremity, severe and insufficiently corrected loss of vision or hearing, severe language difficulties or any other disability that may prevent the participant from cooperating adequately in the trial or that may interfere with neuropsychological test performance.
3. Pre-stroke cognitive impairment (16-item Informant Questionnaire on Cognitive Decline (IQCODE) score ≥ 3.3), preexisting major neurocognitive disorder (e. g., dementia due to Alzheimer's disease, vascular dementia, dementia with Lewy bodies, frontotemporal dementia).
4. Cardiogenic ischemic stroke, atrial fibrillation, or any other conditions that require the intake of anticoagulants.
5. Conditions that require the administration of thrombolytics at day of Screening or Visit 1.
6. Index acute ischemic stroke with hemorrhagic transformation.
7. Intake of traditional Chinese medicines.
8. Major neurological disorder, including intracranial hemorrhage, delirium, Parkinson's disease, brain tumor, alcohol-associated brain damage, infectious CNS disease, epilepsy, recent brain trauma, subdural hematoma, HIV-associated cognitive disorder, Huntington's disease, Pick's disease, Wilson's disease, normal pressure hydrocephalus, hydrocephalus, progressive supra-nuclear palsy, Creutzfeldt-Jakob disease, etc.
9. Major depression or generalized anxiety disorder.
10. Active malignant disease.
11. Alcohol addiction or substance abuse.
12. Known hypersensitivity to Ginkgo biloba, Ginkgo biloba extract or any ingredient of the drug under trial.
13. Any circumstances that prevent the participant to be followed up at the scheduled intervals. Hospitalization of the participant for long-term treatment or nursing home placement for bedside care (assisted living facility residence or stay in a rehabilitation facility is acceptable if the participant is not bedridden and does not need general bedside nursing, and if an informant is available who sees the participant on a regular basis and accompanies him/her to the trial visits).
14. Severe comorbidity with life expectancy < 12 months.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-11-28 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Montreal Cognitive Assessment (MoCA) Total Score | From baseline to Week 26 (Visit 4) and Week 52 (Visit 6)
  The Montreal Cognitive Assessment (MoCA) is a validated screening tool for mild cognitive impairment. It assesses multiple cognitive domains including attention, executive functions, memory, language, visuospatial skills, conceptual thinking, calculation, and orientation. The test takes approximately 10 minutes to administer and is scored out of a maximum of 30 points. The total score is calculated by summing all sub-item scores, with an additional 1 point added for individuals with ≤12 years of education (maximum score remains 30). Higher scores indicate better cognitive performance. A score below 23 for individuals with ≤12 years of education, or below 22 for those with >12 years of education, is considered indicative of cognitive impairment [Wu et al., 2013].
Change in Cognitive Function Using Trail Making Test (TMT) Parts A and B | Change from baseline to Week 26 (Visit 4) and Week 52 (Visit 6)
  The Trail Making Test (TMT) is a neuropsychological assessment that provides information on visual search, scanning, processing speed, mental flexibility, and executive functioning. It consists of two parts. Both parts consist of 25 circles distributed over a sheet of paper. In Part A, the circles are numbered 1 - 25, and the patient should draw lines to connect the numbers in ascending order. In Part B, the circles include both Arabic numerals (1 - 13) and Chinese numerals as in Part A. he test is administered on paper, and participants are instructed to complete the task as quickly and accurately as possible without lifting the pen. Performance is measured in seconds.
Change in Cognitive Processing Speed Using Symbol Digit Modalities Test (SDMT) | Change from baseline to Week 26 (Visit 4) and Week 52 (Visit 6)
  The Symbol Digit Modalities Test (SDMT) is a validated neuropsychological test used to assess cognitive processing speed, attention, and visual-motor coordination. Participants are presented with a series of symbols, each paired with a digit, and are asked to match as many symbols to their corresponding digits as possible within a fixed time period (typically 90 seconds). Performance is measured by the number of correct symbol-digit matches completed (maximum 110). Higher scores indicate better cognitive processing speed and attention
Change in Verbal Fluency Performance Using Verbal Fluency Test (VFT) | Change from baseline to Week 26 (Visit 4) and Week 52 (Visit 6)
  The VFT tests the verbal fluency, the patient is asked to name as many examples of one category, e.g. "fruits", "vegetables", "animal", as possible within one minute. Performance is assessed by counting the number of correct, non-repeated words, along with the number of errors, including incorrect responses and repetitions, which contribute to the total score. Higher scores indicate better verbal fluency and cognitive function.
Change in Clinical Global Impression of Change Using ADCS-CGIC (Alzheimer's Disease Cooperative Study - Clinical Global Impression of Change) | Change from baseline to Week 26 (Visit 4) and Week 52 (Visit 6)
  The Alzheimer's Disease Cooperative Study - Clinical Global Impression of Change (ADCS-CGIC) is a validated clinician-rated instrument used to assess overall change in a participant's cognitive, functional, and behavioral status over time. It is based on a structured interview with both the participant and caregiver, incorporating clinical judgment and observation.
  The ADCS-CGIC uses a 7-point scale to rate change from baseline:
  1. - Marked improvement
  2. - Moderate improvement
  3. - Minimal improvement
  4. - No change
  5. - Minimal worsening
  6. - Moderate worsening
  7. - Marked worsening
  Lower scores indicate improvement, while higher scores reflect deterioration.
Change in Neurological Impairment Using National Institutes of Health Stroke Scale (NIHSS) | Change from Baseline to Week 4 (Visit 1), Week 26 (Visit 4) and Week 52 (Visit 6)
  The National Institutes of Health Stroke Scale (NIHSS) is a standardized tool used to assess the severity of neurological deficits in patients following a stroke. It consists of 11 items evaluating functions such as consciousness, vision, motor skills, sensation, language, and attention. Each item is scored individually, and the total score ranges from 0 to 42, with higher scores indicating more severe neurological impairment. A decrease in score over time reflects improvement in neurological function, while an increase indicates worsening impairment.
Change in Neurological Impairment Using Modified Rankin Scale (mRS) | Change from Baseline to Week 4 (Visit 1), Week 26 (Visit 4) and Week 52 (Visit 6)
  The Modified Rankin Scale (mRS) is a clinical tool for measuring the degree of disability or dependence in daily activities of people who have suffered a stroke. It assesses functional recovery and neurological impairment on a scale ranging from 0 to 6:
  0 - No symptoms at all
  1. - No significant disability despite symptoms; able to carry out all usual duties and activities
  2. - Slight disability; unable to carry out all previous activities but able to look after own affairs without assistance
  3. - Moderate disability; requiring some help, but able to walk without assistance
  4. - Moderately severe disability; unable to walk without assistance, and unable to attend to own bodily needs without assistance
  5. - Severe disability: bedridden, incontinent, and requiring constant nursing care and attention
  6. - Dead
  Lower scores indicate better functional outcomes.
Any new stroke event (ischemic stroke or hemorrhagic stroke) at Week 4, Week 12, Week 26, Week 38 and Week 52. | Week 4, Week 12, Week 26, Week 38 and Week 52

OTHER OUTCOMES:
Incidence and Nature of Adverse Events, Adverse Drug Reactions, and Serious Adverse Events [Safety Assessment] | up to 52 weeks
  Safety will be assessed by documenting the frequency and nature of adverse events (AEs), adverse drug reactions (ADRs), and serious adverse events (SAEs) throughout the entire trial period. Investigators will record the number of participants experiencing each type of event, including details on severity, relationship to study treatment, and outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Petra Klement, Study Director — Dr. Willmar Schwabe GmbH & Co. KG
Locations (12):
- China (12):
  - Baotou Central Hospital, Baotou
  - Tiantan Hospital, Beijing
  - Dalian Lvshunkou District Traditional Chinese Medicine Hospital, Dalian
  - Dalian University Affiliated Xinhua Hospital, Dalian
  - The Second Hospital of Hebei Medical University, Hebei
  - The First Affiliated Hospital of Jiamusi University, Jiamusi
  - Liaocheng People´s Hospital, Liaocheng
  - Liuzhou Workers´ Hospital, Liuchow
  - Second Hospital of Shanxi Medical University, Shanxi
  - Suining Central Hospital, Suining
  - Weifang People´s Hospiztal, Weifang
  - Yantaishan Hospital, Yantai

IPD SHARING:
Plan to Share IPD: No
Due to ethical reasons and in terms of data protection law, raw data cannot be shared

REFERENCES:
- [Background] Wu Y, Wang M, Ren M, Xu W. The effects of educational background on Montreal Cognitive Assessment screening for vascular cognitive impairment, no dementia, caused by ischemic stroke. J Clin Neurosci. 2013 Oct;20(10):1406-10. doi: 10.1016/j.jocn.2012.11.019. Epub 2013 Jul 24. PMID 23891119
- [Background] Liu L, Li Z, Zhou H, Duan W, Huo X, Xu W, Li S, Nie X, Liu H, Liu J, Sun D, Wei Y, Zhang G, Yuan W, Zheng L, Liu J, Wang D, Miao Z, Wang Y. Chinese Stroke Association guidelines for clinical management of ischaemic cerebrovascular diseases: executive summary and 2023 update. Stroke Vasc Neurol. 2023 Dec 29;8(6):e3. doi: 10.1136/svn-2023-002998. PMID 38158224
- [Background] Herrschaft H, Nacu A, Likhachev S, Sholomov I, Hoerr R, Schlaefke S. Ginkgo biloba extract EGb 761(R) in dementia with neuropsychiatric features: a randomised, placebo-controlled trial to confirm the efficacy and safety of a daily dose of 240 mg. J Psychiatr Res. 2012 Jun;46(6):716-23. doi: 10.1016/j.jpsychires.2012.03.003. Epub 2012 Mar 27. PMID 22459264
- [Background] El Husseini N, Katzan IL, Rost NS, Blake ML, Byun E, Pendlebury ST, Aparicio HJ, Marquine MJ, Gottesman RF, Smith EE; American Heart Association Stroke Council; Council on Cardiovascular and Stroke Nursing; Council on Cardiovascular Radiology and Intervention; Council on Hypertension; and Council on Lifestyle and Cardiometabolic Health. Cognitive Impairment After Ischemic and Hemorrhagic Stroke: A Scientific Statement From the American Heart Association/American Stroke Association. Stroke. 2023 Jun;54(6):e272-e291. doi: 10.1161/STR.0000000000000430. Epub 2023 May 1. PMID 37125534
- [Background] Cui M, You T, Zhao Y, Liu R, Guan Y, Liu J, Liu X, Wang X, Dong Q. Ginkgo biloba extract EGb 761(R) improves cognition and overall condition after ischemic stroke: Results from a pilot randomized trial. Front Pharmacol. 2023 Mar 29;14:1147860. doi: 10.3389/fphar.2023.1147860. eCollection 2023. PMID 37063270